CLINICAL TRIAL: NCT01137110
Title: Comparison of Short Duration Levetiracetam to Extended Course Levetiracetam for Seizure Prophylaxis Following Subarachnoid Hemorrhage
Brief Title: Short Duration Levetiracetam to Extended Course for Seizure Prophylaxis After aSAH
Acronym: DOPAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Theresa Human-Murphy, Dr., Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-1717
Record Dates: First submitted 2010-05-28; First posted 2010-06-04 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Hemorrhage; Seizure Prophylaxis; Levetiracetam
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief LEV (Other): Administration of three days of levetiracetam twice daily after SAH
  Interventions: Other: Brief LEV
- Extended LEV (Other): Administration of levetiracetam twice daily after SAH
  Interventions: Other: Extended LEV

INTERVENTIONS:
Other: Brief LEV — Levetiracetam 1000mg BID x 3 days for prophylaxis
  Arms: Brief LEV
Other: Extended LEV — Levetiracetam 1000mg BID for length of hospital stay for prophylaxis
  Arms: Extended LEV

SUMMARY:
Our primary objective is to compare two treatment options for prevention of seizures following a subarachnoid hemorrhage and determine if a short-course regimen of levetiracetam is as efficacious in the prevention of in-hospital seizures when compared to an extended course.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, controlled trial. Patients admitted with spontaneous SAH (and meet enrollment criteria) will be randomized to either levetiracetam 1000 mg twice daily for 3 days or levetiracetam 1000mg twice daily until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age
2. Diagnosis of spontaneous SAH

Exclusion Criteria:

1. SAH secondary to trauma or arteriovenous malformation
2. Early death (defined as death within 3 days of presentation)
3. Known allergy to levetiracetam
4. Know seizure history on chronic AEDs
5. Pregnancy
6. Current incarceration

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Human-Murphy, Principal Investigator — Barnes-Jewish Hospital, Washington University
Locations (1):
- Barnes-jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients enrolled were assigned to a treatment group.
Groups:
- Levetiracetam 1000mg BID for 3 Days: Levetiracetam short course: Levetiracetam 1000mg BID x 3 days
  This cohort will receive three days of Levetiracetam twice daily for seizure prophylaxis. They will be followed for the entire hospital stay for incidence of seizures. If a seizure occurs, the treating physician will treat per usual therapies. Functional status will be assessed at the patients outpatient follow up if available.
- Levetiracetam 1000mg BID x Hospital Stay: Levetiracetam Long course: Levetiracetam 1000mg BID x hospital stay
  This cohort will receive Levetiracetam for the entire length of hospital stay. They will be closely followed for both incidence of seizures as well as adverse effects of the medication. Functional status will be assessed at the patients outpatient follow up if available.
Period: Overall Study
Arm/Group | Levetiracetam 1000mg BID for 3 Days | Levetiracetam 1000mg BID x Hospital Stay
Started | 35 | 49
Completed | 34 | 49
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Brief LEV: 3 days of LEV 1000mg after aSAH
- Extended LEV: LEV for hospital stay after aSAH
- Total: Total of all reporting groups
Arm/Group | Brief LEV | Extended LEV | Total
Number analyzed (Participants) | 35 | 49 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 45 | 77
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 32 | 55
  Male | 12 | 17 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 25 | 39 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: In-hospital Seizures
Description: from admission to In-hospital seizures after aSAH
Time Frame: from hospital admission to hospital discharge
Measure: Count of Participants; unit: Participants
Groups:
- Brief LEV; Extended LEV: In-hospital seizure in patient receiving 3 days of LEV compared to Extended LEV that received LEV for length of hospital stay.
Arm/Group | Brief LEV | Extended LEV
Number analyzed (Participants) | 35 | 49
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: from admission, daily until hosptial discharge.
Groups:
- Brief LEV: ADR requiring discontinuation
- Extended LEV: ADR requiring discontinue
Arm/Group | Brief LEV | Extended LEV
Serious Adverse Events (participants affected / at risk) | 0/35 | 4/49
Other Adverse Events (participants affected / at risk) | 0/35 | 1/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief LEV (N=35) | Extended LEV (N=49)
Sedation (Nervous system disorders) | 0 (0) | 4 (4) — Excessive Sedation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief LEV (N=35) | Extended LEV (N=49)
thrombocytopenia (Immune system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We were unable to achieve our target sample size due to slow enrollment. Secondly, the study was not blinded for the primary outcome which could introduce bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No